CLINICAL TRIAL: NCT03018548
Title: Improvised Explosive Device (IED) Level Blasting of Human Blood With Slosh Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-1087
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- subject blood drawns (Experimental): subjects will have blood drawn which will then be exposed to blast via CO2 cartridge
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — subjects will have blood drawn done. This blood will then be exposed to blasting with CO2 cartridge

SUMMARY:
To monitor changes in indicators of red cell damage such as extracellular hemoglobin, potassium (K-ABL), and lactate dehydrogenase (LD) post blast exposure.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) causes significant morbidity and mortality, accompanied by high related costs. Recent hypotheses concerning the pathophysiology of TBI invoke Strain Shear Theory and Cavitation Theory. The invbestigators propose to test the importance of the latter by directing blast waves into containers that are either partially or completely filled with blood and measuring markers of lysis.

These experiments are designed to better understand the demonstrated effectiveness of mild jugular compression according to the principle of the Queckenstedt Maneuver to reduce the likelihood of TBI by filling up the compliance of the cranial space. A device (C-Collar) is being developed by Q30 Labs, LLC (Q30), to accomplish this effect.

ELIGIBILITY:
Inclusion Criteria:

* • Normal healthy volunteer

  * Able to provide written consent
  * Must be 18 years or older

Exclusion Criteria:

* • Unable to provide written consent

  * Recent penetrating brain trauma (within 6 months)
  * Under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Lysis of blood cells | within 2 hours
  measure the lysis of blood cells exposed to blast from CO2 cartridge

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No